CLINICAL TRIAL: NCT05118230
Title: A Prospective, Observational Study to Assess the Real World Effectiveness of Inclisiran (Leqvio®) in Chinese Adult Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: Study to Assess the Real World Effectiveness of Inclisiran in Chinese Adult Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A1CN01
Record Dates: First submitted 2021-10-26; First posted 2021-11-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Primary Hypercholesterolemia; Mixed Dyslipidemia; Real World Effectiveness; Inclisiran; China
MeSH Terms: interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inclisiran Cohort: patients treated with inclisiran in certain special territories in China
  Interventions: Other: Inclisiran
- SoC Historical Cohort: patients treated with standard of care (SoC) in routine clinical practice from EMR database

INTERVENTIONS:
Other: Inclisiran — Prospective observational study. There is no treatment allocation. Chinese Patients who receive inclisiran in authorized health institutions are eligible to enroll into this study.
  Groups: Inclisiran Cohort

SUMMARY:
This is a multi-center, prospective, comparative and non-interventional cohort study involving two cohorts, one cohort (Inclisiran Cohort) of patients treated with inclisiran in certain special territories in China (eg. Bo'ao Pilot Zone) and the other cohort (SoC Historical Cohort) of patients treated with standard of care (SoC) in routine clinical practice from EMR database.

DETAILED DESCRIPTION:
This study will utilize real-world data from EMR database to serve as the 'external control'.The purpose of this study is to compare the effectiveness of inclisiran as an add-on therapy (or monotherapy in statin-intolerant cases) in real-world settings, with current SoC in a matched historical cohort of patients who receive SoC in EMR database.

The patients in Inclisiran Cohort will received inclisiran injection (300 mg s.c.) under the guidance of physicians, and based on the approved label, which recommends a second dose on 90 days after the first injection, and then followed by injections every 6 months afterwards until the end of study (EOS). However, the treatment decision and exact visit timepoint will be purely decided by physicians and patients.

ELIGIBILITY:
Inclusion Criteria:

Inclisiran Cohort Patients eligible for inclusion in this study must meet all of the following criteria.

1. Confirmed diagnosis of primary hypercholesterolemia or mixed dyslipidemia
2. Age ≥ 18 years at baseline
3. Initiated treatment with inclisiran according to the decision of both physician and patient
4. Signed informed consent(s) must be obtained prior to participation in the study

SoC Historical Cohort Patients eligible for inclusion in this study must meet all of the following criteria.

1. Confirmed diagnosis of primary hypercholesterolemia or mixed dyslipidemia, with which reference to LDL-C > 70 mg/dL (1.8 mmol/L)
2. Age ≥ 18 years
3. Compliance with the standard lipid-lowering therapy, which is defined as a change from prior lipid-lowering therapy to an optimal lipid-lowering regimen, with the date of compliance with standard lipid-lowering therapy after January 1, 2017 as the index date
4. With available LDL-C test at baseline, which is defined as the closest LDL-C test to the index date within 6 months prior to the index date
5. With available LDL-C test on D90 (90±60 days) or D330 (330±90 days) after the index date

Exclusion Criteria:

Inclisiran Cohort Patients meeting any of the following criteria are not eligible for inclusion in this study.

1. Treatment with monoclonal antibodies directed towards PCSK9 within 90 days before first visit (V1)
2. Severe hepatic impairment (Child-Pugh class C)
3. Severe renal impairment (eGFR ≤ 30 mL/min), and/or on hemodialysis
4. Participation in any cardiovascular clinical trial, concurrent or within the last 30 days of the baseline
5. Females who are pregnant or nursing, or who are preparing for pregnancy
6. Hypersensitivity to the active substance or to any of the excipients of inclisiran solution

SoC Historical Cohort Patients meeting any of the following criteria are not eligible for inclusion in this study.

1. Treatment with monoclonal antibodies directed towards PCSK9 during research period
2. Severe hepatic impairment (Child-Pugh class C)
3. Severe renal impairment, (eGFR ≤ 30 mL/min), and/or on hemodialysis
4. Participation in any cardiovascular clinical trial during research period
5. Females who are pregnant or nursing during research period

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who receive inclisiran in authorized health institutions and eligible patients from EMR database.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Percentage change in LDL-C from baseline | Baseline, Day 330
  To assess the real-world effectiveness of inclisiran plus SoC in reducing LDL-C in reference to a matched historical cohort of SoC.

SECONDARY OUTCOMES:
Change in LDL-C from baseline | Baseline, Day 90, Day 150, Day 270, Day 330,Day 450 and Day 510
  Percentage and absolute change will be provided
Change in total cholesterol, HDL-C, Lp(a) and triglycerides from baseline | Baseline, Day 90, Day 150, Day 270, Day 330, Day 450 and Day 510
  Percentage and absolute change will be provided
Proportion of patients discontinuing from inclisiran during the study and the reasons for treatment discontinuation if available | Day 150
  If the planned dose is missed for more than 3 months, the patient is considered as discontinuation.
Proportion of patients with treatment switch and reinitiation during the study | Day 150
  * Switch: defined as patient starts monoclonal antibody treatment directed towards PCSK9. Switching date is defined as the date of the first claim of the new therapy.
  * Reinitiation: defined as patient previously discontinues inclisiran > 9 months (from last dose received), and then reinitiates inclisiran.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- China (2):
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Qionghai, Hainan

IPD SHARING:
Plan to Share IPD: No